CLINICAL TRIAL: NCT06761963
Title: Chronic Effect of Whole-body Electrical Stimulation in COPD Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Santa Casa de Porto Alegre (Other)
Responsible Party: Principal Investigator, Jociane Schardong, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WBES_COPD_2
Record Dates: First submitted 2024-11-04; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole-body electrical stimulation (Experimental): Performed with calibrated Miha Bodytec equipment, with electrodes on the quadriceps, hamstrings, glutes, biceps, triceps, pectorals, abdomen, trapezius, latissimus dorsi, and quadratus lumborum. A symmetrical biphasic current, 400µs pulse width, 75Hz frequency will be used. Sixteen sessions will occur twice weekly for eight weeks. In weeks 1-2, contractions last five seconds with 10 seconds rest, for 16 minutes (64 contractions). In weeks 3-5, contractions remain five seconds with five seconds rest, also lasting 16 minutes (96 contractions). In weeks 6-8, contractions/rest stay at five seconds each, lasting 20 minutes (120 contractions). Initial isometric positions familiarize the patient with stimulation, followed by squats, biceps/triceps exercises with a proprioception stick, abdominal exercises, step-up exercises, and aerobic activities (bike/treadmill) to conclude each session.
  Interventions: Other: Whole-body electrical stimulation
- Rehabilitation (Other): There will be 16 sessions, twice a week, on alternate days, for eight weeks. It will consist of muscle strengthening exercises, using weights, ankle weights and weight training equipment. Squats, biceps and triceps exercises (with weights), knee flexion and extension (equipment with weights) and stretching will be performed. At the end of each session, patients will do aerobic exercise (bicycle or treadmill).
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Whole-body electrical stimulation — Performed using Miha Bodytec equipment, properly calibrated, with electrodes on the quadriceps, hamstrings, glutes, biceps, triceps, pectorals, abdomen, trapezius, latissimus dorsi and quadratus lumborum muscles.
  Arms: whole-body electrical stimulation
Other: Rehabilitation — Pulmonary rehabilitation program.
  Arms: Rehabilitation

SUMMARY:
Randomized clinical trial. Patients with chronic obstructive pulmonary disease (COPD) GOLD III or IV will undergo 16 sessions of Whole-body Electrical Stimulation (WB-EMS) or pulmonary rehabilitation (PR), twice a week. WB-EMS will be performed in association with squats, biceps and triceps exercises, climbing up and down a step, and abdominal exercises. There will be a progression in the number of muscle contractions after the fourth (from 64 to 96) and tenth sessions (96 to 120). PR will consist of upper and lower limb strengthening exercises. Both groups will perform aerobic exercise (essential component of the pulmonary rehabilitation program). Peripheral muscle strength (dynamometry), respiratory muscle strength (maximum inspiratory and expiratory pressure), muscle thickness (ultrasound), functional capacity (6MWT), quality of life (Saint George's Respiratory Questionnaire), inflammatory profile (PCR, IL-6 e IL-10, TNFα), oxidative stress (protein oxidation, superoxide dismutase and catalase, total hydrogen sulfides, dichlorofluorescein diacetate) will be assessed before and after the 16 sessions.

DETAILED DESCRIPTION:
Patients with chronic obstructive pulmonary disease (COPD) will undergo a 16-session whole-body electrical stimulation (WB-EMS) protocol or a pulmonary rehabilitation program, twice a week, for eight weeks. The Miha Bodytec equipment will be properly calibrated, with electrodes on the quadriceps, hamstrings, glutes, biceps, triceps, pectorals, abdomen, trapezius, latissimus dorsi and quadratus lumborum muscles. Symmetrical pulsed biphasic current will be used, pulse width of 400 µs, frequency of 75 Hz. In the first two weeks, the contraction time will be five seconds and the rest time will be 10 seconds, the session will last 16 minutes, resulting in 64 muscle contractions. In weeks 3, 4 and 5, the contraction time will be five seconds and the rest time will be five seconds, the session will last 16 minutes, resulting in 96 muscle contractions. In weeks 6, 7 and 8, the contraction time will be five seconds and the rest time will be five seconds. The session will last 20 minutes, resulting in 120 muscle contractions. During the first two minutes of stimulation, the patient will remain in isometric position to familiarize themselves with the electrical current. After that, a series of squats, biceps and triceps exercises (using a proprioception stick), abdominal exercises and climbing up and down a step will be performed. At the end of each session, patients will do aerobic exercise (bicycle or treadmill). Pulmonary rehabilitation will consist of muscle strengthening exercises, using weights, ankle weights and weight training equipment. Squats, biceps and triceps exercises (with weights), knee flexion and extension (equipment with weights) and stretching will be performed. At the end of each session, patients will do aerobic exercise (bicycle or treadmill). Peripheral muscle strength (dynamometry), respiratory muscle strength (maximum inspiratory and expiratory pressure), muscle thickness (ultrasound), functional capacity (6MWT), quality of life (Saint George's Respiratory Questionnaire), inflammatory profile (PCR, IL-6 e IL-10, TNFα), oxidative stress (protein oxidation, superoxide dismutase and catalase, total hydrogen sulfides, dichlorofluorescein diacetate) will be assessed before and after the 16 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD GOLD 3 and 4;
* Age between 18 and 80 years;
* Ability to ambulate.

Exclusion Criteria:

* Cognitive dysfunction that prevents assessments from being carried out, as well as inability to understand and sign the informed consent form (ICF);
* Intolerance to the electrostimulator and/or change in skin sensitivity;
* Patients with stroke sequelae;
* Recent acute myocardial infarction (two months);
* Uncontrolled hypertension;
* New York Heart Association grade IV heart failure or decompensated;
* Unstable angina or arrhythmia;
* Peripheral vascular changes in lower limbs such as deep vein thrombosis;
* Disabling osteoarticular or musculoskeletal disease;
* Uncontrolled diabetes (glycemia > 300mg/dL);
* Patients with cancer and/or undergoing cancer treatment;
* Patients with systemic lupus erythematosus or other autoimmune disease;
* Artificial cardiac pacemaker;
* Epilepsy;
* Hemophilia;
* Liver and kidney diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Peripheral muscle strength | Baseline
  Peripheral muscle strength will be assessed by maximum isometric strength of the knee extensor, elbow flexor and palmar flexor muscles using a hand-held dynamometer
Peripheral muscle strength | Two months
  Peripheral muscle strength will be assessed by maximum isometric strength of the knee extensor, elbow flexor and palmar flexor muscles using a hand-held dynamometer

SECONDARY OUTCOMES:
Maximum inspiratory pressure | Baseline
  Maximum inspiratory pressure will be assessed by manovacuometry.
Maximum inspiratory pressure | Two months
  Maximum inspiratory pressure will be assessed by manovacuometry.
Maximum expiratory pressure | Baseline
  Maximum expiratory pressure will be assessed by manovacuometry.
Maximum expiratory pressure | Two months
  Maximum expiratory pressure will be assessed by manovacuometry.
Muscle thickness | Baseline
  Muscle thickness will be assessed by the thickness of the quadriceps, biceps and abdominal muscles using ultrasound
Muscle thickness | Two months
  Muscle thickness will be assessed by the thickness of the quadriceps, biceps and abdominal muscles using ultrasound
Functional capacity | Baseline
  Functional capacity will be assessed by the Six-minute walk test
Functional capacity | Two months
  Functional capacity will be assessed by the Six-minute walk test
Quality of life | Baseline
  Quality of life will be assessed by the Saint George's Respiratory Questionnaire. Scores range from 0 to 100, with higher scores indicating more limitations
Quality of life | Two months
  Quality of life will be assessed by the Saint George's Respiratory Questionnaire. Scores range from 0 to 100, with higher scores indicating more limitations
Inflammatory profile | Baseline
  The inflammatory profile will be assessed by the levels of PCR, IL-6 e IL-10, TNFα
Inflammatory profile | Two months
  The inflammatory profile will be assessed by the levels of PCR, IL-6 e IL-10, TNFα
Oxidative stress | Baseline
  The oxidative stress will be assessed by the measurement of protein oxidation, superoxide dismutase and catalase, total hydrogen sulfides, dichlorofluorescein diacetate
Oxidative stress | Two months
  The oxidative stress will be assessed by the measurement of protein oxidation, superoxide dismutase and catalase, total hydrogen sulfides, dichlorofluorescein diacetate

IPD SHARING:
Plan to Share IPD: No